CLINICAL TRIAL: NCT01272960
Title: Randomized, Open-label, Controlled Trial of Immediate Postpartum Versus Interval Insertion of Mirena to Increase the Usage at 6 Months After Delivery
Brief Title: Mirena Intrauterine System Timing of Insertion: A Randomized Controlled Trial
Acronym: MISTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SFP4-13
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Postpartum Period
Keywords: Contraception; Postnatal care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interval Insertion (Active Comparator): Will receive Mirena at 4-8 weeks post-partum after vaginal delivery.
  Interventions: Device: Interval Insertion
- Post-Placental Mirena Insertion (Experimental): Will receive Mirena insertion within 10 minutes of delivery of placenta
  Interventions: Device: Post-Placenta Mirena Insertion

INTERVENTIONS:
Device: Post-Placenta Mirena Insertion — Mirena(R) intrauterine device will be inserted within 10 minutes of delivery of the placenta
  Arms: Post-Placental Mirena Insertion
Device: Interval Insertion — Insertion of Mirena 4-8 weeks post partum after vaginal delivery
  Arms: Interval Insertion

SUMMARY:
In order to determine the timing of LNG-IUS insertion that results in a greater proportion of women using the LNG-IUS at 6-months post-partum, we will perform a randomized control trial of interval versus immediate post-placenta insertion. Women will be enrolled at 36-weeks gestation and greater. At the time of vaginal delivery, women will be randomized to receive either immediate post-placenta insertion of the LNG-IUS or routine insertion at 4-8 weeks post-partum. All patients will return at 4-6 weeks post-insertion and 6 months post-partum to confirm correct position of the LNG-IUS. The primary outcome of this sub-study is the number of LNG-IUS in the correct position at 6-months. Secondary outcomes include assessing the safety of post-placental LNG-IUS insertion and difference in acceptability and symptoms experienced by participants. This is a sub-study of the Contraceptive Choice Project, a prospective cohort study that aims to improve the use of long-acting contraception by removing financial barriers which has already enrolled over 5,000 patients. Association of this study with CHOICE offers unique advantages including infrastructure to support subject recruitment, retention and completion of follow-up as well as covering the cost of LNG-IUS devices.

We hypothesize that, despite higher expulsion rates, women randomized to receive the LNG-IUS immediately after placenta delivery will have higher rates of LNG-IUS continuation due to poor rates of follow up in the interval insertion group. This is likely to be particularly noticeable in our patient population, which is largely uninsured with poor access to healthcare. Further, typical symptoms of LNG-IUS insertion include bleeding and cramping, which may be disguised by the post-partum period. Published reports of immediate post-placenta insertion focus on expulsion rates and do not report on symptoms and satisfaction rates.

ELIGIBILITY:
Inclusion Criteria:

* 14-45 years
* Vaginal Delivery at Barnes-Jewish Hospital
* Sexually active with male partner
* No tubal ligation/hysterectomy
* Not currently using contraception
* Desire reversible contraception
* Reside in St. Louis City/County
* Requests Mirena(R) intrauterine device for contraception

Exclusion Criteria:

* Allergy to Mirena(R) system
* Cesarean delivery
* Cervical cancer, breast cancer
* Active liver disease
* Untreated cervicitis
* Uterine anomaly/fibroids preventing Mirena(R) placement
* Delivery <36 weeks
* Chorioamnionitis
* Prolonged rupture of membranes (>18 hours)

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorie M Harper, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Finer LB, Henshaw SK. Disparities in rates of unintended pregnancy in the United States, 1994 and 2001. Perspect Sex Reprod Health. 2006 Jun;38(2):90-6. doi: 10.1363/psrh.38.090.06. PMID 16772190
- [Background] Gillett PG, Lee NH, Yuzpe AA, Cerskus I. A comparison of the efficacy and acceptability of the Copper-7 intrauterine device following immediate or delayed insertion after first-trimester therapeutic abortion. Fertil Steril. 1980 Aug;34(2):121-4. doi: 10.1016/s0015-0282(16)44893-4. No abstract available. PMID 7409230
- [Background] Sivin I, Stern J. Health during prolonged use of levonorgestrel 20 micrograms/d and the copper TCu 380Ag intrauterine contraceptive devices: a multicenter study. International Committee for Contraception Research (ICCR). Fertil Steril. 1994 Jan;61(1):70-7. doi: 10.1016/s0015-0282(16)56455-3. PMID 8293847
- [Background] Comparative multicentre trial of three IUDs inserted immediately following delivery of the placenta. Contraception. 1980 Jul;22(1):9-18. doi: 10.1016/0010-7824(80)90112-2. PMID 7418410
- [Background] Thiery M, Van Kets H, Van der Pas H. Immediate post-placental IUD insertion: the expulsion problem. Contraception. 1985 Apr;31(4):331-49. doi: 10.1016/0010-7824(85)90002-2. PMID 4006467
- [Background] Morrison C, Waszak C, Katz K, Diabate F, Mate EM. Clinical outcomes of two early postpartum IUD insertion programs in Africa. Contraception. 1996 Jan;53(1):17-21. doi: 10.1016/0010-7824(95)00254-5. PMID 8631184
- [Background] Xu JX, Reusche C, Burdan A. Immediate postplacental insertion of the intrauterine device: a review of Chinese and the world's experiences. Adv Contracept. 1994 Mar;10(1):71-82. doi: 10.1007/BF01986532. PMID 8030457
- [Background] Zhou SW, Chi IC. Immediate postpartum IUD insertions in a Chinese hospital--a two year follow-up. Int J Gynaecol Obstet. 1991 Jun;35(2):157-64. doi: 10.1016/0020-7292(91)90820-u. PMID 1680090
- [Background] Eroglu K, Akkuzu G, Vural G, Dilbaz B, Akin A, Taskin L, Haberal A. Comparison of efficacy and complications of IUD insertion in immediate postplacental/early postpartum period with interval period: 1 year follow-up. Contraception. 2006 Nov;74(5):376-81. doi: 10.1016/j.contraception.2006.07.003. Epub 2006 Sep 15. PMID 17046378
- [Background] Chen BA, Reeves MF, Hayes JL, Hohmann HL, Perriera LK, Creinin MD. Postplacental or delayed insertion of the levonorgestrel intrauterine device after vaginal delivery: a randomized controlled trial. Obstet Gynecol. 2010 Nov;116(5):1079-87. doi: 10.1097/AOG.0b013e3181f73fac. PMID 20966692

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 53 participants were enrolled but only 29 randomized.
Groups:
- Interval Insertion: Will receive Mirena at 4-8 weeks post-partum after vaginal delivery.
  Post-Placenta Mirena Insertion: Mirena(R) intrauterine device will be inserted within 10 minutes of delivery of the placenta
Period: Overall Study
Arm/Group | Interval Insertion | Post-Placental Mirena Insertion
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Interval Insertion: 14 subjects received Mirena at 4-8 weeks post-partum after vaginal delivery.
- Post-Placental Mirena Insertion: 15 received Mirena insertion within 10 minutes of delivery of placenta
- Total: Total of all reporting groups
Arm/Group | Interval Insertion | Post-Placental Mirena Insertion | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (4.6) | 26.9 (4.2) | 26.6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29
Number of pregnancies at viable gestational age [Number; unit: Pregnancies] | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mirena in Place
Description: Proportion of women in each arm with Mirena in place at 6 months
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Post Placental Mirena Insertion | Interval Insertion
Number analyzed (Participants) | 15 | 14
participants | 10 | 3

2. Secondary Outcome: Mirena Expulsion
Description: The percentage of patients with post-placental placement of Mirena who experience an expulsion
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Interval Insertion | Post-Placental Mirena Insertion
Number analyzed (Participants) | 14 | 15
participants | 0 | 0

3. Secondary Outcome: Uterine Perforation
Description: The proportion of patients in each arm who experience a uterine perforation
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Interval Insertion | Post-Placental Mirena Insertion
Number analyzed (Participants) | 14 | 15
participants | 0 | 0

4. Secondary Outcome: Intrauterine Infection
Description: The proportion of patients in each arm who experience an intrauterine infection (endometritis, pelvic inflammatory disease)
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Interval Insertion | Post-Placental Mirena Insertion
Number analyzed (Participants) | 14 | 15
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Interval Insertion | Post Placental Mirena Insertion
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interval Insertion (N=14) | Post Placental Mirena Insertion (N=15)
Infection (Infections and infestations) | 0 (0) | 1 (1) — One LNG-IUS was removed in the immediate insertion group and not replaced due to a systemic Group B streptococcus infection diagnosed within 6-weeks post-partum.

LIMITATIONS AND CAVEATS:
Inability to recruit and randomize our target sample size, to detect rare adverse events that may be associated with immediate insertion, women randomized to immediate insertion were more likely to return for their 6-month string check visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No